CLINICAL TRIAL: NCT06819605
Title: Neoadjuvant Therapy With Dabrafenib and Trametinib Followed by Curettage/Fenestration Surgery Versus Up-front Curettage and Fenestration Surgery in BRAF V600E Mutated Ameloblastoma: A Randomized Controlled Clinical Trial
Brief Title: Neoadjuvant Therapy With Conservative Surgery vs. Up-front Conservative Surgery for BRAF V600E-Mutated Ameloblastoma
Acronym: NETCAM-RCT
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NETCAM_2025CT; SH9H-2024-T470-1 (Other: Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine Ethics Committee)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Ameloblastoma
Keywords: Ameloblastoma; Neoadjuvant therapy; Curettage and fenestration surgery; Recurrence - free survival rate; BRAF V600E
MeSH Terms: conditions — Ameloblastoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Curettage and fenestration surgery alone
- Neoadjuvant group (Experimental): Neoadjuvant therapy chemotherapy before curettage and fenestration surgery
  Interventions: Drug: Dabrafenib and trametinib (combination)

INTERVENTIONS:
Drug: Dabrafenib and trametinib (combination) — This clinical study investigates the combination of Dabrafenib (2 mg once daily for adults; 0.025 mg/kg/day for children ≥12 years, orally once daily) and Trametinib (2 mg once daily for adults; 0.025 mg/kg/day for children ≥12 years, orally once daily) as a treatment for [specific condition]. The treatment will be administered until disease progression or intolerable toxicities occur. Both medications should be taken at least 1 hour before or 2 hours after a meal, at the same time each day. If a dose is missed, it should be taken within 12 hours of the scheduled time. If less than 12 hours remain before the next dose, the missed dose should not be taken. Both medications should be taken in combination with the scheduled dose of Dabrafenib at either morning or evening and must not be chewed or crushed.
  Each treatment cycle lasts 30 days. At the end of each cycle, follow-up assessments will include clinical examination, laboratory tests to evaluate drug safety, and imaging studies to a
  Arms: Neoadjuvant group

SUMMARY:
Ameloblastoma is the most common benign odontogenic tumor, characterized by high local invasiveness and a high recurrence rate. Currently, surgical treatment is the standard treatment modality. The main surgical approaches include radical resection represented by local extended resection (with a safety margin of more than 2 cm) and conservative procedures represented by curettage and fenestration. Although radical resection can effectively treat the disease, it often leads to severe jaw bone defects and even disrupts the continuity of the jaw bone. However, the conservative procedures have a recurrence rate of approximately 40%.

This study aims to reduce the recurrence rate of conservative procedures by using neoadjuvant therapy with dabrafenib combined with trametinib, and to reduce surgical trauma while improving the radical cure effect. The endpoints of this study are the 3-year and 5-year recurrence rates, as well as the effectiveness and safety of the neoadjuvant therapy.

DETAILED DESCRIPTION:
The primary endpoints are the 3-year and 5-year recurrence - free survival rates after neoadjuvant therapy followed by curettage and fenestration surgery. The secondary endpoints are the radiological response, pathological response, and safety of the neoadjuvant therapy with dabrafenib combined with trametinib.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years.
* Pathologically confirmed diagnosis of solid or cystic ameloblastic tumors, or recurrent unicystic ameloblastic tumors.
* Presence of BRAF V600E mutation confirmed by next-generation sequencing (NGS) in tumor tissue.
* Requires mandible resection at initial diagnosis (limited to segmental mandibulectomy, subtotal maxillectomy, or total maxillectomy).
* No distant metastasis or malignancy.
* ECOG performance status of 0-1.
* Willing to undergo surgical treatment after neoadjuvant therapy.
* No significant contraindications to MEK inhibitors or BRAF inhibitors.
* Adequate organ function as defined by the following standards: a) Hematologic criteria: WBC ≥ 4.0 × 10^9/L, ANC ≥ 1.5 × 10^9/L, PLT ≥ 100 × 10^9/L, Hb ≥ 90 g/L (no blood transfusion or blood products within the past 14 days, no G-CSF or other hematopoietic growth factors used to correct). b) Biochemical criteria: Serum albumin ≥ 3.0 g/dL (30 g/L), TBIL ≤ 1.5 × ULN, ALT, AST ≤ 2.5 × ULN, BUN and CRE ≤ 1.5 × ULN or estimated creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula). c) Normal coagulation function: Defined as INR or PT ≤ 1.5 × ULN; for patients on anticoagulant therapy, PT within the therapeutic range for the anticoagulant drug.
* Women of childbearing potential must have used reliable contraception, undergone a pregnancy test within 7 days prior to enrollment with a negative result, and be willing to continue using effective contraception during the study and for 16 weeks after the last dose of Trametinib combined with Dabrafenib. Male participants with female partners of childbearing potential should use effective contraception during the study and for 16 weeks after the last dose of Trametinib combined with Dabrafenib.

Exclusion Criteria:

* Previous treatment with Dabrafenib, Trametinib, or any other BRAF inhibitors or MEK inhibitors.
* Presence of active autoimmune disease. Subjects with stable autoimmune conditions not requiring systemic immunosuppressive therapy are allowed, such as: type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, and skin conditions that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia).
* Congenital or acquired immunodeficiency (e.g., HIV infection), active hepatitis B (HBV-DNA ≥ 10^4 copies/ml), or hepatitis C (positive HCV antibodies with HCV RNA above the detection threshold of the testing method).
* Known allergy to the study drugs or any of their excipients; or a history of severe allergic reaction to other monoclonal antibodies or targeted therapies.
* History of myocardial infarction, severe/uncontrolled angina, NYHA class ≥2 heart failure, clinically significant supraventricular or ventricular arrhythmias, or symptomatic congestive heart failure within 6 months prior to enrollment.
* Receipt of a live vaccine within 4 weeks prior to first dose of study drug. Seasonal influenza vaccines are allowed if inactivated and injected, but live attenuated influenza vaccines (e.g., nasal spray) are not allowed.
* Known history of organ transplantation or hematopoietic stem cell transplantation.
* Known history of substance abuse or drug addiction.
* Pregnant or breastfeeding women.
* Diagnosis of any other malignancy within 5 years prior to study entry, except for cured localized skin basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, ductal carcinoma in situ of the breast, papillary thyroid carcinoma, and benign tumors.
* Presence of other serious physical or mental health conditions, or laboratory abnormalities that may increase the risk of participating in the study or interfere with the study results, as determined by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence - free survival rates | Up to 5 years
  To evaluate the recurrence-free survival after neoadjuvant therapy with dabrafenib and trametinib, followed by curettage and fenestration surgery.

SECONDARY OUTCOMES:
Radiological response | 3 months
  The radiological response to neoadjuvant therapy with Dabrafenib and Trametinib in patients with ameloblastoma will be assessed through three-dimensional volumetric imaging (e.g., CT scans with 3D reconstruction) at predefined intervals. Tumor volume changes, as determined by 3D reconstruction, will be used to evaluate the radiological response.
Pathological response | 4 months
  The pathological response to neoadjuvant therapy with Dabrafenib and Trametinib in patients with ameloblastoma will be assessed through post-treatment surgical specimens.
AEs will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 1 year
  The safety of neoadjuvant therapy with Dabrafenib and Trametinib in patients with ameloblastoma will be assessed through monitoring adverse events (AEs). AEs will be recorded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, and graded based on severity (Grade 1 to Grade 5) and their relationship to the study drugs.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grynberg S, Vered M, Shapira-Frommer R, Asher N, Ben-Betzalel G, Stoff R, Steinberg Y, Amariglio N, Greenberg G, Barshack I, Toren A, Yahalom R, Schachter J, Rechavi G, Hirschhorn A, Abebe Campino G. Neoadjuvant BRAF-targeted therapy for ameloblastoma of the mandible: an organ preservation approach. J Natl Cancer Inst. 2024 Apr 5;116(4):539-546. doi: 10.1093/jnci/djad232. PMID 37966914
- [Result] Gasparro R, Giordano F, Campana MD, Aliberti A, Landolfo E, Dolce P, Sammartino G, di Lauro AE. The Effect of Conservative vs. Radical Treatment of Ameloblastoma on Recurrence Rate and Quality of Life: An Umbrella Review. J Clin Med. 2024 Sep 9;13(17):5339. doi: 10.3390/jcm13175339. PMID 39274556